CLINICAL TRIAL: NCT01935609
Title: Evaluation of a Skill-Building, Supportive, and Educational Intervention for Couples (a Research Project Within the Traumatic Brain Injury Model System Grant)
Brief Title: Evaluation of a Skill-Building, Supportive, and Educational Intervention for Couples
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: HM14736; H133A120031 (Other Grant/Funding Number: NIDILRR)
Record Dates: First submitted 2013-08-21; First posted 2013-09-05 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Traumatic Brain Injury; Acquired Brain Injury
Keywords: traumatic brain injury; acquired brain injury
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Injuries

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Couples counseling (Experimental): Intervention to promote couples' adjustment (TCI) - The TCI was developed based upon considerable clinical experience and research review. The TCI is a structured approach to helping couples after brain injury address issues related to relationship quality and emotional well-being. The TCI is implemented in five or six (optional parenting session) session. Each session is in-person and lasts for 120 minutes.
  Interventions: Behavioral: Couples counseling
- Waitlist Control (No Intervention): Couples are randomly assigned to the treatment group or waitlist control (WLC) group. Couples will complete the study measures on 2 occasions, 5 weeks apart. In fairness, WLC couples will then be offered the opportunity to participate in the intervention.

INTERVENTIONS:
Behavioral: Couples counseling — Intervention to promote couples' adjustment (TCI) - The TCI was developed based upon considerable clinical experience and research review. The TCI is a structured approach to helping couples after brain injury address issues related to relationship quality and emotional well-being. The TCI is implemented in five or six (optional parenting session) session. Each session is in-person and lasts for 120 minutes.
  Arms: Couples counseling

SUMMARY:
1. To evaluate the efficacy of a structured outpatient couples intervention program (Therapeutic Couples Intervention, TCI) on couples' marital quality after acquired brain injury (ABI).
2. To assess the impact of the TCI on the emotional well-being of persons with ABI and their partners.
3. To ascertain the impact of the TCI on caregiver burden and unmet needs as reported by partners of persons with ABI.
4. To examine the extent to which treatment benefits for survivors and their caregiving partners are sustained in the longer-term.

DETAILED DESCRIPTION:
Much of the research on acquired brain injury (ABI) has focused on survivors, especially functional and neurobehavioral outcomes. In recent years, researchers have begun to develop and evaluate interventions designed to improve whole family functioning. Studies have demonstrated that intervention can increase survivors' and family members' problem solving skills, met needs, emotional adjustment, and perceptions about the quality of rehabilitation services.

Research suggests at least one of every three survivors is in a martial or coupled relationship at the time of injury. The literature examining postinjury marital breakdown has yielded widely varying results with estimates of breakdown rates ranging from 15%-78%. Whereas early studies suggested a majority of marriages ended in divorce, more recent studies have indicated that marital breakdown rates for people with brain injury are substantially lower than the general population. At the same time, research has generated concern that while many people remain together the quality of the relationship is sorely diminished.

There is little doubt that healthy marriages and intimate relationships are important elements of our society. Further, research in other medical disciplines has proven the positive impact marital quality has on marital stability, emotional well-being, caregiver burden, and family needs. Existing study has similarly established the sustained benefits of promoting marital quality through intervention. Given the documented adverse impacts of brain injury, there is a clear need for effective interventions to improve and maintain the quality of coupled relationships.

To improve couples' relationship quality after ABI, and to target emotional well-being and caregiver burden, VCU researchers developed a curriculum-based program for couples (Therapeutic Couples Intervention, TCI). The study addresses issues and challenges commonly confronting couples after brain injury. Relationship quality is a primary focus of the study with the perceptions of both partners analyzed, allowing an understanding of individual viewpoints and those of the couple as a whole. Objectives include:

1. to evaluate the efficacy of a structured outpatient couples intervention program (TCI) on couples' marital quality
2. to assess the impact of the TCI on the emotional well-being of persons with ABI and their partners
3. to ascertain the impact of the TCI on caregiver burden and unmet needs as reported by partners of persons with ABI
4. to examine the extent to which treatment benefits for survivors and their caregiving partners are sustained in the longer-term

ELIGIBILITY:
Inclusion Criteria:

* partners and persons with ABI who are at least three months post-injury or post-diagnosis
* ABI is defined as damage to brain tissue caused by aneurysm, brain abscess, stroke, anoxia, or non-progressive brain tumor, or an external mechanical force as evidenced by: loss of consciousness due to brain trauma, post-traumatic amnesia (PTA), skull fracture, or objective neurological findings that can be reasonably attributed to ABI on physical examination or mental status examination.
* a "partner" is defined as a person described by the individual with the injury as a spouse, partner, or significant other
* able to understand and provide consent

Exclusion Criteria:

* active substance abusers (e.g., intoxicated at arrival to intake)
* at imminent risk of psychiatric hospitalization
* in imminent danger of hurting themselves or others
* individuals without a partner

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2013-03; Primary Completion 2016-09-28 (Actual); Study Completion 2016-09-28 (Actual)

PRIMARY OUTCOMES:
Revised Dyadic Adjustment Scale (RDAS) | Change from Baseline to Post-Treatment (5-6 weeks after Baseline)
  Couples' relationship quality will be measured using the Revised Dyadic Adjustment Scale (RDAS), an improved version of the Dyadic Adjustment Scale (DAS). The RDAS has 14 items which are rated using a Likert type scale with values ranging from 0-5 or 0-4. Total scores range from 0-69 with higher values indicating greater marital quality. Scores < 48 are indicative of a distressed relationship. The RDAS has been found to be successful at distinguishing between distressed and non-distressed couples and is sensitive to treatment effects. Examples of items include, "Do you ever regret that you married or moved in together?," "Do you and your mate engage in outside interests together?," and "How often do you and your partner have a good conversation?" As done in other studies using the R-DAS, the present investigation will rely on the mean Total Score, incorporating Total Scores from each member of the couple.

SECONDARY OUTCOMES:
Brief Symptom Inventory-18 (BSI) | Change from Baseline to Post-Treatment (5-6 weeks after Baseline)
  The Brief Symptom Inventory-18 (BSI-18) is an 18 item self-report instrument designed to quantify psychological distress in the general population. Increasingly, the measure has been used to quantify individuals and family members' distress after ABI. The instrument is a psychometrically sound, abbreviated version of the SCL-90-R. Frequency ratings for items in three primary symptom dimensions are added to yield scores for Somatization, Depression, and Anxiety. The Global Severity Index (GSI) reflects the sum of scores for the three symptom dimensions. T-scores for each dimension and the GSI are calculated based on community norms. GSI scores, reflecting overall distress levels, will be used in the present investigation.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey S Kreutzer, PhD, Principal Investigator — Professor, Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Graham KM, Kreutzer JS, Marwitz JH, Sima AP, Hsu NH. Can a couples' intervention reduce unmet needs and caregiver burden after brain injury? Rehabil Psychol. 2020 Nov;65(4):409-417. doi: 10.1037/rep0000300. Epub 2019 Dec 19. PMID 31855018